CLINICAL TRIAL: NCT02582307
Title: Hyoscine Hydrobromide (Buscopan) Versus Acetaminophen for Acute Abdominal Pain in Children: A Randomized Controlled Trial
Brief Title: Buscopan Versus Acetaminophen for Acute Abdominal Pain in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 107243
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Abdomen, Acute; Children
MeSH Terms: conditions — Abdomen, Acute | interventions — Acetaminophen; Analgesics; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyoscine butylbromide (Experimental): Hyoscine butylbromide 10mg oral single dose
  Interventions: Drug: Hyoscine butylbromide, Analgesics, Non-Narcotic
- Acetaminophen (Active Comparator): Acetaminophen 15mg/kg oral single dose (maximum 1000mg)
  Interventions: Drug: Acetaminophen, Analgesics, Non-Narcotic

INTERVENTIONS:
Drug: Acetaminophen, Analgesics, Non-Narcotic — Oral single dose
  Other Names: Tylenol
  Arms: Acetaminophen
Drug: Hyoscine butylbromide, Analgesics, Non-Narcotic — Oral single dose
  Other Names: Buscopan
  Arms: Hyoscine butylbromide

SUMMARY:
There is ample evidence that pain in children is under recognized and under treated. This is especially true for acute abdominal pain, a common complaint in the paediatric emergency department. Clinicians often fear that analgesia will obscure the diagnosis of a potentially surgical condition. As a result, acute abdominal pain goes untreated in many children, as there is no standard of care. Hyoscine N-butylbromide (Buscopan) has been used successfully in adults and children for pain associated with urinary tract infections and kidney stones for over 60 years. However, no study has explored its usefulness in relieving acute abdominal pain in children. The objectives of this study are to investigate to what degree Buscopan is effective in relieving abdominal pain in children compared to acetaminophen.

DETAILED DESCRIPTION:
Acute abdominal pain is a common complaint among paediatric patients visiting the emergency department (ED). Functional abdominal pain is not associated with any surgical or infectious etiology and is a frequent cause of painful abdominal cramps. Although functional abdominal pain is not life-threatening, it has significant impact on quality of life, functional outcomes, and patient satisfaction. It is a major source of school and work absence, loss of sleep, and extracurricular impairment. Despite this, analgesia has traditionally been withheld from patients with acute abdominal pain. The reasons behind this are likely two-fold. First, there is good evidence that clinicians fear that analgesia will mask signs of an underlying surgical pathology such as appendicitis. There is no current published literature that supports this practice. In fact, recent evidence has found that providing analgesia to children does not obscure signs of an acute surgical abdomen nor lead to clinically significant differences in negative outcomes. Second, there is no standard of care specifying the best analgesic options for treating abdominal pain in children in the post-codeine era. Although acetaminophen, ibuprofen, ketorolac, buscopan, and almagel/viscous lidocaine are frequently used agents in the ED, evidence for their benefit in children with functional abdominal pain is lacking. As a predictable result, most patients who present with abdominal pain fail to experience pain relief at discharge. The importance of providing optimal pain treatment is echoed by several national and international level policy statements. In addition to the World Health Organization (WHO)'s mandate that adequate pain treatment should be a fundamental human right, the American Academy of Pediatrics (AAP) has reaffirmed its position that adequate analgesia be provided for children. Furthermore, literature supports that providing analgesia improves patient care, caregiver satisfaction, and the therapeutic relationship. Antispasmodics are commonly used agents to treat abdominal cramping. Hyoscine butylbromide (HBB), trade name: Buscopan, is an anticholinergic agent that when orally administered, does not cross the blood brain barrier and has minimal systemic absorption. Therefore, it inhibits bowel motility without central nervous system or peripheral side effects. This antispasmodic has been used in clinical practice for over 60 years and specifically has been on the market since 1952 for the treatment of abdominal cramps. It is widely available around the world as both a prescription drug and an over the counter medication in many industrialized countries. It has also been used safely in neonates and children. As hyoscine butylbromide is barely absorbed, it is generally well tolerated. In the two large-scale studies of almost 1200 patients that compared HBB with placebo (and paracetamol), there was no significant difference in adverse events between the two groups, including those commonly associated with anticholinergics, such as nausea, constipation, dry mouth, blurred vision, tachycardia and urinary retention. Moreover, these adverse events not only occurred at a low incidence (less than or equal to 1.5%) but were also usually mild and self-limiting. In abdominal cramping and pain associated with irritable bowel syndrome, systematic reviews have had conflicting results with regards to analgesic efficacy, primarily because of small sample sizes and less rigorous designs. Muller-Krampe et al. conducted a prospective cohort of over 200 children with both acute and chronic abdominal spasms and compared the effectiveness of oral HBB 10 mg to a homeopathic preparation. HBB demonstrated comparative improvements to the homeopathic preparation with respect to pain, sleep disturbance, eating and drinking, and crying. Over 90% of patients in both groups reported good tolerability and there were no adverse events. Although HBB is used widely for abdominal pain in children and anecdotal evidence suggests it is efficacious, no paediatric clinical trial to date has explored its efficacy in the ED setting. The investigators hypothesize that HBB will have superior efficacy to the most commonly used agent, acetaminophen for acute abdominal pain in children. If HBB is found to be an effective analgesic in children with acute abdominal pain, it could provide a therapeutic option for a common, painful condition for which there is currently very little to offer.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 8-17 years presenting to the paediatric ED with:

  1. A chief complaint of colicky abdominal pain AND
  2. Pain score of at least 4/10 on the Faces Pain Scale - Revised AND
  3. A presumed non-surgical etiology

Exclusion Criteria:

1. Prior abdominal surgery
2. Concomitant use of other anticholinergic medication including but not limited to tricyclic antidepressants, antihistamines, benztropine mesylate
3. Signs and symptoms consistent with a bowel obstruction
4. Peritoneal signs
5. Suspected previous hypersensitivity reaction to either acetaminophen or HBB
6. Suspected appendicitis
7. History of abdominal trauma within 48 hours of presentation
8. Unstable vital signs
9. History of bowel obstruction
10. Myasthenia gravis
11. Fever (aural temperature > 38.2 C)
12. Chronic liver disease
13. Persistent vomiting despite administration of oral anti-emetic
14. Symptoms and signs consistent with a urinary tract infection
15. Symptoms and signs consistent with a toxin ingestion
16. Symptoms and signs consistent with gynecological or gonadal pathology
17. Symptoms and signs consistent with vasoocclusive crisis in a patient with a hemoglobinopathy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Analgesic Efficacy | 80 minutes post-intervention
  Pain severity on a 100 mm Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Analgesic Efficacy | 15 minutes post-intervention
  Pain severity on Faces Pain Scale - Revised and VAS
Analgesic Efficacy | 30 minutes post-intervention
  Pain severity on Faces Pain Scale - Revised and VAS
Analgesic Efficacy | 45 minutes post-intervention
  Pain severity on Faces Pain Scale - Revised and VAS
Analgesic Efficacy | 60 minutes post-intervention
  Pain severity on Faces Pain Scale - Revised and VAS
Need for Rescue Analgesia | 80 minutes post-intervention
  Frequency of rescue analgesia
Time to Analgesia | 80 minutes post-intervention
  Time to Achieve 20% Reduction in Faces Pain Score - Revised from time 0
Adequacy of Sedation | 80 minutes post-intervention
  Proportion of participants that achieve a pain score < 30 mm on the VAS
Adverse Effects | 80 minutes post-intervention
  Frequency of Adverse Effects
Caregiver Satisfaction | 80 minutes post-intervention
  Satisfaction scores on 5-Item Likert Scale
Return visits | 72 hours post discharge
  Proportion of participants with return visits for surgical pathology

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MD, Principal Investigator — Western University Health
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poonai N, Kumar K, Coriolano K, Thompson G, Brahmbhatt S, Dzongowski E, Stevens H, Gupta P, Miller M, Elsie S, Ashok D, Joubert G, Lim R, Butter A, Ali S. Hyoscine butylbromide versus acetaminophen for nonspecific colicky abdominal pain in children: a randomized controlled trial. CMAJ. 2020 Nov 30;192(48):E1612-E1619. doi: 10.1503/cmaj.201055. PMID 33257343